CLINICAL TRIAL: NCT03661138
Title: A Phase 3 Randomized, Multicenter, Double-Blind Study to Evaluate the Safety of Upadacitinib in Combination With Topical Corticosteroids in Adolescent and Adult Subjects in Japan With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate Safety of Upadacitinib in Combination With Topical Corticosteroids in Adolescent and Adult Participants With Moderate to Severe Atopic Dermatitis
Acronym: Rising Up
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M17-377; 2022-002777-29 (EudraCT Number)
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Atopic Dermatitis
Keywords: Upadacitinib; Topical Corticosteroids; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — upadacitinib; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A (Experimental): Upadacitinib Dose A is administered once daily along with Topical Corticosteroids (TCS).
  Interventions: Drug: Upadacitinib; Drug: Topical Corticosteroids (TCS)
- Arm B (Experimental): Upadacitinib Dose B is administered once daily along with Topical Corticosteroids (TCS).
  Interventions: Drug: Upadacitinib; Drug: Topical Corticosteroids (TCS)
- Arm C (Experimental): Placebo administered once daily and TCS followed by Upadacitinib Dose A once daily along with TCS.
  Interventions: Drug: Upadacitinib; Drug: Placebo for upadacitinib; Drug: Topical Corticosteroids (TCS)
- Arm D (Experimental): Placebo administered once daily and TCS followed by Upadacitinib Dose B once daily along with TCS.
  Interventions: Drug: Upadacitinib; Drug: Placebo for upadacitinib; Drug: Topical Corticosteroids (TCS)

INTERVENTIONS:
Drug: Upadacitinib — Upadacitinib is administered orally.
  Other Names: ABT-494
Drug: Placebo for upadacitinib — Placebo is administered orally.
  Arms: Arm C; Arm D
Drug: Topical Corticosteroids (TCS) — It is administered concomitantly with upadacitinib or placebo.

SUMMARY:
The objective of this study is to assess the safety of upadacitinib combined with topical corticosteroids (TCS) in adolescent and adult participants in Japan with moderate to severe atopic dermatitis (AD) who are candidates for systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Active moderate to severe atopic dermatitis defined by Eczema Area and Severity Index (EASI), Investigator's Global Assessment (IGA), Body surface area (BSA), and pruritus.
* Candidate for systemic therapy or have recently required systemic therapy for atopic dermatitis.
* Able to tolerate topical corticosteroids for atopic dermatitis lesions.

Exclusion Criteria:

* Prior exposure to any Janus kinase (JAK) inhibitor.
* Unable or unwilling to discontinue current atopic dermatitis (AD) treatments prior to the study.
* Requirement of prohibited medications during the study.
* Female participant who is pregnant, breastfeeding, or considering pregnancy during the study.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2018-10-27 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing adverse events | Up to 141 Weeks
  Adverse events are defined as those that began or worsened in severity after the first dose of study drug but within 30 days after the last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (43):
- Japan (43):
  - Ichinomiya Municipal Hospital /ID# 205942, Ichinomiya-shi, Aichi-ken
  - Central Clinic /ID# 206558, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 207566, Nagoya, Aichi-ken
  - Yasumoto Dermatology Clinic /ID# 206480, Chikushino-shi, Fukuoka
  - Kiryu Dermatology Clinic /ID# 206044, Fukuoka, Fukuoka
  - Medical Corporation Matsuo Clinic /ID# 207323, Fukuoka, Fukuoka
  - Matsuda Tomoko Dermatological Clinic /ID# 206288, Fukuoka, Fukuoka
  - Higuchi Dermatology Urology Clinic /ID# 206287, Kasuga-shi, Fukuoka
  - Central Japan International Medical Center /ID# 205684, Minokamo-shi, Gifu
  - Kiryu Kosei General Hospital /ID# 206155, Kiryu-shi, Gunma
  - Gunma University Hospital /ID# 207016, Maebashi, Gunma
  - Fukuyama City Hospital /ID# 206761, Fukuyama-shi, Hiroshima
  - Asahikawa Medical University Hospital /ID# 206521, Asahikawa-shi, Hokkaido
  - Medical Corporation Kato Dermatology Clinic /ID# 206561, Sapporo, Hokkaido
  - Kitago Dermatology Clinic /ID# 207025, Sapporo, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 206519, Sapporo, Hokkaido
  - Kansai Rosai Hospital /ID# 205918, Amagasaki-shi, Hyōgo
  - Hyogo Prefectural Amagasaki General Medical Center /ID# 206974, Amagasaki-shi, Hyōgo
  - Kobe University Hospital /ID# 206200, Kobe, Hyōgo
  - Tokai University Hospital /ID# 206657, Isehara-shi, Kanagawa
  - Medical corporation Kojunkai Kosugi Dermatology Clinic /ID# 206766, Kawasaki-shi, Kanagawa
  - Nippon Medical School Musashi Kosugi Hospital /ID# 206656, Kawasaki-shi, Kanagawa
  - Yokohama Rosai Hospital /ID# 206648, Yokohama, Kanagawa
  - Suizenji Dermatology Clinic /ID# 205871, Kumamoto, Kumamoto
  - Nagasaki University Hospital /ID# 206118, Nagasaki, Nagasaki
  - Nagaoka Red Cross Hospital /ID# 209817, Nagaoka-shi, Niigata
  - Isonokami dermatological clinic /ID# 206923, Daito-shi, Osaka
  - Medical corporation Kojinkai Yoshioka Dermatology Clinic /ID# 209704, Neyagawa, Osaka
  - Shizuoka General Hospital /ID# 207122, Shizuoka, Shizuoka
  - Mildix Skin Clinic /ID# 206829, Adachi-ku, Tokyo
  - Yaesu Nihonbashi Skin Clinic /ID# 207125, Chuo-ku, Tokyo
  - Fukuwa clinic /ID# 206760, Chuo-ku, Tokyo
  - Hosono Clinic /ID# 205953, Chuo-ku, Tokyo
  - Nihon University Itabashi Hospital /ID# 206186, Itabashi-ku, Tokyo
  - Mita Dermatology /ID# 206694, Minato-ku, Tokyo
  - Medical Corporation Jitai-kai Nakano Dermatology Clinic /ID# 206882, Nakano-ku, Tokyo
  - Matsuyama Dermatology /ID# 205998, Nakano-ku, Tokyo
  - Miu Skin Clinic /ID# 206911, Ōta-ku, Tokyo
  - Tokyo Rosai Hospital /ID# 205809, Ōta-ku, Tokyo
  - Tampopo Dermatology Clinic /ID# 207013, Ōta-ku, Tokyo
  - Naoko Dermatology Clinic /ID# 205334, Setagaya-ku, Tokyo
  - Tachikawa Dermatology Clinic /ID# 206996, Tachikawa-shi, Tokyo
  - Toyama Prefectural Central Hospital /ID# 206286, Toyama, Toyama

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Katoh N, Ikeda M, Ohya Y, Murota H, Hu X, Liu J, Niiyama H, Sasaki T, Raymundo EM, Saeki H. Safety and Efficacy of Upadacitinib for Atopic Dermatitis in Japan: Analysis of the 3-Year Phase 3 Rising Up Study. Dermatol Ther (Heidelb). 2024 Jan;14(1):213-232. doi: 10.1007/s13555-023-01071-2. Epub 2023 Dec 21. PMID 38127188
- [Derived] Hayashi N, Ikeda M, Liu J, Raymundo E, Liu Y, Sasaki T, Yamasaki K. Acne Among Japanese Patients with Atopic Dermatitis Receiving Upadacitinib in the Phase 3 Rising Up Study. Dermatol Ther (Heidelb). 2023 Aug;13(8):1817-1830. doi: 10.1007/s13555-023-00961-9. Epub 2023 Jun 25. PMID 37356075
- [Derived] Katoh N, Ohya Y, Murota H, Ikeda M, Hu X, Ikeda K, Liu J, Sasaki T, Raymundo EM, Teixeira HD, Saeki H. Safety and Efficacy of Upadacitinib for Atopic Dermatitis in Japan: 2-Year Interim Results from the Phase 3 Rising Up Study. Dermatol Ther (Heidelb). 2023 Jan;13(1):221-234. doi: 10.1007/s13555-022-00842-7. Epub 2022 Nov 19. PMID 36401761
- [Derived] Tanaka T, Sasaki T, Ikeda K, Liu J, Tenorio AR, Ohya Y. Growth analysis among adolescents with moderate-to-severe atopic dermatitis receiving upadacitinib in combination with topical corticosteroids in Japan: A case study series from a phase 3, randomized, controlled trial (Rising Up). World Allergy Organ J. 2022 Sep 13;15(9):100678. doi: 10.1016/j.waojou.2022.100678. eCollection 2022 Sep. PMID 36185549
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M17-377&Latitude=&Longitude=&LocationName=#additional-resources-section